CLINICAL TRIAL: NCT07193537
Title: Virtual Reality Exercises Versus Motor Control Training on Cervical Proprioception in Symptomatic Forward Head Posture
Brief Title: Virtual Reality Exercises Versus Motor Control Training in Symptomatic Forward Head Posture
Acronym: VRexercises
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Nabil Abdelmageed, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: exercises on symptomatic FHP
Record Dates: First submitted 2025-09-24; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Symptomatic Forward Head Posture
Keywords: pain
MeSH Terms: conditions — Pain | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: Virtual reality systems have been used in assessments and treatments in the field of rehabilitation .
  Motor control training motor control training of deep neck flexors with pressure biofeedback is an effective intervention for improving pain intensity and disability in patients with neck pain and preferable to strength-endurance training of cervical muscles . Scapular stabilization exercise can help improve the head posture and pain in the patients with neck pain and forward head posture.
  conventional treatment in form of Posture correction (chin tuck exercise) and Stretching exercises
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality exercises (Experimental): Thirty one subjects will receive virtual reality exercises by VR Training using Xbox Kinect for four weeks .
  Interventions: Other: Virtual reality exercises
- Motor control training (Experimental): Motor control training for four weeks
  Interventions: Other: Motor control training
- conventional treatment (Active Comparator): conventional treatment for four weeks in form of posture correction and stretching exercises
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: Virtual reality exercises — Thirty one subjects will receive virtual reality exercises by VR Training using Xbox Kinect. The Kinect sensor is an infrared camera that can recognize the positions and motions of the player without the need for special controller. The console controls the various games .For the VR training, the Xbox Kinect, console, and monitor will set up in a dedicated space. The patient will placed 1.5-2 m away from the Kinect sensor. Before the start of the training session, the research assistant adjusted the position of the sensor while the patient is sitting to ensure optimal position and motion capture, and loaded games into the system. After the setup is completed, the research assistant demonstrated games included in the Kinect adventure
  Arms: Virtual reality exercises
Other: Motor control training — Thirty one subjects will receive motor control training two times a week for eight weeks in form of deep cervical flexors strengthening using pressure biofeedback unit (craniocervical flexor exercise) :Pressure biofeedback unit will be used to perform Cranio-cervical flexor muscle training. Through which an endurance and isometric exercise for DNFs in progressive range positions will be performed each session, the PBU's air bag will be positioned below the occiput, and the inflatable cuff pressure sensor will be inflated to a baseline of 20 mmHg. Participants will instruct to target five pressure levels between 22 and 30 mmHg by nodding. scapular exercises .With patient in prone position, pillow under the chest and upper limb in varying degree of shoulder abduction, the participant lifts the hand toward the ceiling while retracting the scapula
  Arms: Motor control training
Other: conventional treatment — Thirty one subjects will receive conventional treatment for 3 times per week for 4 weeks. Conventional treatment will include the following:
  1-Posture correction (chin tuck exercise) Stand with the upper back against the wall, with the feet shoulder-width apart. Tuck the chin in and hold for 5 seconds 10 repetitions .Return to the starting position and repeat a number of times. This can help stretch the muscles in the upper neck 2. Stretching exercise: Self-stretching exercise for most common tight muscles. These muscles include upper trapezius (by contralateral side bending), levator scapulae (flexion, contralateral side bending and rotation) and sternocleidomastoid muscle (slight flexion with ipsilateral side bending and rotation). Each position should be maintained for 30 seconds and repeated for 3 times.
  Arms: conventional treatment

SUMMARY:
This study will be conducted to Compare between virtual reality exercises versus motor control training on cervical proprioception in symptomatic forward head posture

DETAILED DESCRIPTION:
Various occupations require people to maintain a static position for long periods that causes continuous contractions of the head and neck muscle.The poor posture leads to pain and deformity such as forward head posture.Virtual reality exercises(VRE) have been more commonly considered for the improvement of pain , functional ability, and muscular strength.Motor control training (MCT) re-establish the activation pattern of neck muscles and have proven to be effective in improving motor function of deep cervical muscles, reducing discomfort and impairment in patient with FHP and neck pain. 93 subjects from both sexes will participate in the study with CVA less than 50º.Group A:31 subjects will receive virtual reality exercises by VR Training using Xbox Kinect

.Group B: 31 subjects will receive motor control training Group C: 31 subjects will receive conventional treatment in form of (Posture correction (chin tuck exercise)and Stretching exercises .

ELIGIBILITY:
Inclusion Criteria:

1. Ninety three subjects from both sexes will participate in the study with CVA less than 50º.
2. Subject's age ranged from 18-30 years old, with Body Mass Index (BMI) less than 30Kg/m2. .
3. Subjects having neck pain more than 6 weeks .
4. Neck disability index (NDI) value less than 24 (mild to moderate disability scores on NDI)

Exclusion Criteria:

1-Individuals with a recent history of neck or back surgery. 2- Individuals with recent history of trauma or fracture. 3- Individuals with congenital disorders 4- Individuals with any psychiatric diseases

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
cervical propioception | up to four weeks
  Cervical proprioception will be assessed using CROM .
Craniovertebral angle (CVA) | up to four weeks
  Photogrammetric method will be used to assess CVA

SECONDARY OUTCOMES:
pain intensity | up to four weeks
  Visual Analogue Scale (VAS) to assess pain intensity
Neck function | up to four weeks
  Arabic version of neck disability index will be used to assess neck function
Deep neck flexors endurance | up to four weeks
  Pressure Biofeedback Unit (PBU, Chattanooga, TN, USA) will be used to assess endurance